CLINICAL TRIAL: NCT00231738
Title: Effect of Eicosapentaenoic Acid (EPA) on Major Cardiovascular Events in Hypercholesterolemic Patients: the Japan EPA Lipid Intervention Study (JELIS)
Brief Title: Protective Effect of EPA on Cardiovascular Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kobe University (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MYokoyama - 001
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2005-10

CONDITIONS: Myocardial Infarction, Unstable Angina Pectoris, Sudden Cardiac Death, Stroke, Peripheral Artery Disease
Keywords: Eicosapentaenoic acid; Coronary artery disease
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Death, Sudden, Cardiac; Stroke; Peripheral Arterial Disease; Coronary Artery Disease

INTERVENTIONS:
Drug: Eicosapentaenoic acid ethyl ester(EPADEL Capsule 300 TM)

SUMMARY:
The purpose of this study was to test the hypothesis that the long-term use of highly (>98%) purified EPA, in addition to HMG-CoA reductase inhibitor (statin), would be more effective than statin alone in preventing cardiovascular events in Japanese patients with hypercholesterolemia.

DETAILED DESCRIPTION:
Epidemiological studies from many countries including Finland, Italy, Japan, and The Netherlands have suggested that an increased intake of dietary fish or fish oil rich in the long-chain polyunsaturated n-3 fatty acids (PUFAs), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), is inversely related to the risk of atherothrombotic diseases, in particular coronary artery disease (CAD).

Results of many prospective observational cohort studies have found that diets rich in marine PUFAs may be protective against major cardiovascular events, including mortality from CAD, total cardiovascular death, all-cause mortality, and nonfatal myocardial infarction. To date, only a few studies have examined the effects of purified n-3 PUFA preparations in human subjects for short observation periods. The principle aim of the current study is to test the hypothesis that the long-term use of highly purified EPA(eicosapentaenoic acid: 1800mg/day), in addition to HMG-CoA reductase inhibitor, is effective in preventing cardiovascular events in Japanese patients with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants had a total cholesterol level of ≧250mg/dL(6.5m mol/L) at baseline.
* Hyperlipidemic patients with serum total cholesterol of 250mg/dL or more. (Measurement of serum total cholesterol)
* Serum total cholesterol should be measured twice at interval of 2-4weeks. A single measurement is acceptable if the cholesterol is measured by blood collection at fasting under strict compliance with dietary advice after withdrawal of the antihyperlipemic drug.
* (Wash Out) The wash out period of 4weeks (8 weeks for probucol) is necessary in patients under treatment with antihyperlipemic drug. However, if treatment with the antihyperlipemic drug was started within 6 months of the initiation of the study, the patient can participate in the study without the washout period.

Exclusion Criteria:

* Acute myocardial infarction occurring within last 6 months
* Unstable angina pectoris
* A history or complication of serious heart disease(severe arrhythmia, heart failure, cardiac myopathy, valvular disease, congenital disease, etc.)
* Receiving cardiovascular reconstruction within last 6 months
* Cerebrovascular disorders occurring within last 6 months
* Complication of serious hepatic disease or renal disease
* Malignant tumor
* Uncontrollable diabetes
* Hyperlipidemia arising from the following disease: Nephrotic syndrome, hypothyroidism, Cushing's syndrome, secondary hyperlipidemia due to other disease
* Hyperlipidemia due to some drugs such as steroid hormone
* Hemorrhage(hemophilia, capillary fragility, gastrointestinal ulcer, urinary tract hemorrhage, hemoptysis, vitreous hemorrhage, etc.)
* Hemorrhagic diathesis
* Hypersensitivity to the study drug formulation
* Patients intending to undergo surgery
* Patients judged to be inappropriate by the physician in charge

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18000
Dates: Start 1996-11; Study Completion 2004-11

PRIMARY OUTCOMES:
Major coronary events (sudden cardiac death, fatal and nonfatal myocardial infarction, unstable angina pectoris including hospitalization for ischemic episodes,events of angioplasty/ stenting or coronary artery bypass grafting)

SECONDARY OUTCOMES:
All-cause mortality
Stroke
Peripheral artery disease; and
Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiro Yokoyama, MD, PhD., Principal Investigator
Locations (1):
- Kobe University Graduate School of Medicine Cardiovascular and Respiratory Medicine Division, Department of Internal Medicine, Kobe, Hyōgo, Japan

REFERENCES:
- [Background] Yokoyama M, Origasa H; JELIS Investigators. Effects of eicosapentaenoic acid on cardiovascular events in Japanese patients with hypercholesterolemia: rationale, design, and baseline characteristics of the Japan EPA Lipid Intervention Study (JELIS). Am Heart J. 2003 Oct;146(4):613-20. doi: 10.1016/S0002-8703(03)00367-3. PMID 14564313
- [Derived] Ishikawa Y, Yokoyama M, Saito Y, Matsuzaki M, Origasa H, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K, Matsuzawa Y; JELIS Investigators. Preventive effects of eicosapentaenoic acid on coronary artery disease in patients with peripheral artery disease. Circ J. 2010 Jul;74(7):1451-7. doi: 10.1253/circj.cj-09-0520. Epub 2010 May 18. PMID 20484828
- [Derived] Origasa H, Yokoyama M, Matsuzaki M, Saito Y, Matsuzawa Y; JELIS Investigators. Clinical importance of adherence to treatment with eicosapentaenoic acid by patients with hypercholesterolemia. Circ J. 2010 Mar;74(3):510-7. doi: 10.1253/circj.cj-09-0746. Epub 2010 Feb 9. PMID 20145342
- [Derived] Oikawa S, Yokoyama M, Origasa H, Matsuzaki M, Matsuzawa Y, Saito Y, Ishikawa Y, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; JELIS Investigators, Japan. Suppressive effect of EPA on the incidence of coronary events in hypercholesterolemia with impaired glucose metabolism: Sub-analysis of the Japan EPA Lipid Intervention Study (JELIS). Atherosclerosis. 2009 Oct;206(2):535-9. doi: 10.1016/j.atherosclerosis.2009.03.029. Epub 2009 Apr 5. PMID 19447387
- [Derived] Matsuzaki M, Yokoyama M, Saito Y, Origasa H, Ishikawa Y, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K, Matsuzawa Y; JELIS Investigators. Incremental effects of eicosapentaenoic acid on cardiovascular events in statin-treated patients with coronary artery disease. Circ J. 2009 Jul;73(7):1283-90. doi: 10.1253/circj.cj-08-1197. Epub 2009 May 8. PMID 19423946
- [Derived] Saito Y, Yokoyama M, Origasa H, Matsuzaki M, Matsuzawa Y, Ishikawa Y, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; JELIS Investigators, Japan. Effects of EPA on coronary artery disease in hypercholesterolemic patients with multiple risk factors: sub-analysis of primary prevention cases from the Japan EPA Lipid Intervention Study (JELIS). Atherosclerosis. 2008 Sep;200(1):135-40. doi: 10.1016/j.atherosclerosis.2008.06.003. Epub 2008 Jun 19. PMID 18667204
- [Derived] Tanaka K, Ishikawa Y, Yokoyama M, Origasa H, Matsuzaki M, Saito Y, Matsuzawa Y, Sasaki J, Oikawa S, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; JELIS Investigators, Japan. Reduction in the recurrence of stroke by eicosapentaenoic acid for hypercholesterolemic patients: subanalysis of the JELIS trial. Stroke. 2008 Jul;39(7):2052-8. doi: 10.1161/STROKEAHA.107.509455. Epub 2008 May 1. PMID 18451347
- [Derived] Yokoyama M, Origasa H, Matsuzaki M, Matsuzawa Y, Saito Y, Ishikawa Y, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; Japan EPA lipid intervention study (JELIS) Investigators. Effects of eicosapentaenoic acid on major coronary events in hypercholesterolaemic patients (JELIS): a randomised open-label, blinded endpoint analysis. Lancet. 2007 Mar 31;369(9567):1090-8. doi: 10.1016/S0140-6736(07)60527-3. PMID 17398308